CLINICAL TRIAL: NCT03313115
Title: Sleep/Wake Protocol Implementation to Improve Sleep Quality and Reduce Delirium in a Surgical and Cardiovascular Intensive Care Unit
Brief Title: Sleep/Wake Protocol Implementation to Improve Sleep Quality in the ICU
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Other Study IDs: 104449
Record Dates: First submitted 2017-10-11; First posted 2017-10-18 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2020-02

CONDITIONS: Sleep Deprivation; Delirium
MeSH Terms: conditions — Sleep Deprivation; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Sleep/Wake Protocol Implementation: No implementation of the sleep/wake protocol. A subset of participants in this group will have light and sound levels in the room recorded.
- Sleep/Wake Protocol Implementation: The sleep/wake protocol will be implemented. A subset of participants in this group will also have light and sound levels in the room recorded.
  Interventions: Behavioral: Sleep/Wake Protocol

INTERVENTIONS:
Behavioral: Sleep/Wake Protocol — Day RN observes if completed per pt: no caffeine after 3 pm, encourage activities to prevent napping (chart % day spent napping), Lights on blinds/door open, Reasonable effort for some noise in room, Eye glasses hearing aids applied, Chair position/mobility at least 2x30 minutes.
  Night RN observe if completed per pt: Appropriate pain control, Optimize room temp, Warm bath before 2200, TV off by 2200, Prevent extra alarms after 2200, Close room curtain by 2200, Dim room lights by 2200, Family out by 2200, Door half/fully closed after 2200, # RN interruptions after 2200, Offer eye mask/ear plugs, Meds administered for sleep (dilaudid, fentanyl oxycodone, haldol, quetiapine, propofol, melatonin, or other), Dim hallway lights by 2200, Nurses station quiet
  Groups: Sleep/Wake Protocol Implementation

SUMMARY:
The purpose of this study is to analyze a multi-component sleep/wake protocol for optimization of environmental factors (noise, light, nursing activities) as well as non-environmental factors (pain, mechanical support devices, procedures) to improve quality of sleep and decrease incidence of ICU delirium in the Cardiovascular and Surgical ICU (CVICU/SICU).

DETAILED DESCRIPTION:
Fifty-percent of ICU patient sleep hours occur during the day in short bouts which decreases overall sleep quality. Approximately 47-87% of critically ill patients in the ICU experience an episode of delirium, which can result in changes in cognition, longer hospital stay, and physiologic consequences. Research suggests that both patients and staff members can identify environmental factors, such as noise, light, and nursing activities, as well as non-environmental factors such as mechanical devices, procedures, and medications as contributing factors to lack of sleep. However, both nursing staff and providers may underestimate the intensity of the perceived noise in the ICU. This includes those frequent nighttime interruptions, of environmental and non-environmental origins, which can cause fragmented sleep. Providers and nurses are aware of the factors contributing to sleep deprivation, but they may "lower prioritization of patient sleep [as a] tradeoff [for] current standard of care."

Studies have shown that sleep deprivation in critically ill patients can lead to changes in patient cognition, increased hospital and ICU length of stay, and physiologic consequences. These consequences are influenced from patient clinical status as well as modifiable risk factors. One study identified that barriers to the optimization of sleep include patient disease severity, mechanical ventilation, sedation, noise, light, and nurse-patient interaction. It identified a possible association between lack of sleep and cognition with additional consequences of longer mechanical ventilator time, and cardiovascular, pulmonary, and immune system dysfunctions.

Implementation of a protocol directed at optimizing environmental and non-environmental factors has been shown to improve patients' perceived and actual quality of sleep as well as a reduction in ICU delirium.

Another study studied sleep and delirium in a medical ICU after implementation of sleep-promoting interventions. Interventions aimed at reducing light, noise, nursing interruptions, and sedating medications were applied in a three-part process. Patients were surveyed using the Richards-Campbell Sleep Questionnaire and delirium was measured by delirium/coma-free days. Post-interventions resulted in an increase in delirium/coma-free days and an improvement in the amount of perceived noise.

One research group implemented a similar bundle that was aimed at improvement of sleep and delirium in both medical and surgical ICU patients. Their efforts were directed towards reduction in environmental factors as well as avoidance of sedating medications and long mechanical ventilator times. The Richards-Campbell Sleep Questionnaire was used to survey patients on quality of sleep and the Confusion Assessment Method for the ICU was measured daily for incidence of delirium. They found that patients' perceived quality of sleep increased with decreased daytime sleepiness as well as reductions in noise, light, and nursing interventions. Furthermore, they found that implementation of this bundle led to a decrease in length of delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Admitted to the cardiovascular or surgical ICU

Exclusion Criteria:

* Patient acuity does not allow nighttime activities to be grouped (i.e., patient requires frequent bedside care throughout the night, as evaluated by registered nurse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be drawn from those admitted into the Cardiovascular or Surgical Intensive Care Units at the University of Utah University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-14 (Actual)

PRIMARY OUTCOMES:
Incidence of ICU delirium | Two times daily until ICU discharge (up to 4 months)
  Participants will be evaluated for delirium using the Confusion Assessment Method for the ICU (CAM-ICU)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tonna, MD, FAAEM, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Beltrami FG, Nguyen XL, Pichereau C, Maury E, Fleury B, Fagondes S. Sleep in the intensive care unit. J Bras Pneumol. 2015 Nov-Dec;41(6):539-46. doi: 10.1590/S1806-37562015000000056. PMID 26785964
- [Background] Bihari S, Doug McEvoy R, Matheson E, Kim S, Woodman RJ, Bersten AD. Factors affecting sleep quality of patients in intensive care unit. J Clin Sleep Med. 2012 Jun 15;8(3):301-7. doi: 10.5664/jcsm.1920. PMID 22701388
- [Background] Cavallazzi R, Saad M, Marik PE. Delirium in the ICU: an overview. Ann Intensive Care. 2012 Dec 27;2(1):49. doi: 10.1186/2110-5820-2-49. PMID 23270646
- [Background] Giusti GD, Tuteri D, Giontella M. Nursing Interactions With Intensive Care Unit Patients Affected by Sleep Deprivation: An Observational Study. Dimens Crit Care Nurs. 2016 May-Jun;35(3):154-9. doi: 10.1097/DCC.0000000000000177. PMID 27043401
- [Background] Hata RK, Han L, Slade J, Miyahira A, Passion C, Ghows M, Izumi K, Yu M. Promoting sleep in the adult surgical intensive care unit patients to prevent delirium. Nurs Clin North Am. 2014 Sep;49(3):383-97. doi: 10.1016/j.cnur.2014.05.012. PMID 25155537
- [Background] Hopper K, Fried TR, Pisani MA. Health care worker attitudes and identified barriers to patient sleep in the medical intensive care unit. Heart Lung. 2015 Mar-Apr;44(2):95-9. doi: 10.1016/j.hrtlng.2015.01.011. Epub 2015 Feb 14. PMID 25686516
- [Background] Kamdar BB, Needham DM, Collop NA. Sleep deprivation in critical illness: its role in physical and psychological recovery. J Intensive Care Med. 2012 Mar-Apr;27(2):97-111. doi: 10.1177/0885066610394322. Epub 2011 Jan 10. PMID 21220271
- [Background] Kamdar BB, King LM, Collop NA, Sakamuri S, Colantuoni E, Neufeld KJ, Bienvenu OJ, Rowden AM, Touradji P, Brower RG, Needham DM. The effect of a quality improvement intervention on perceived sleep quality and cognition in a medical ICU. Crit Care Med. 2013 Mar;41(3):800-9. doi: 10.1097/CCM.0b013e3182746442. PMID 23314584
- [Background] Patel J, Baldwin J, Bunting P, Laha S. The effect of a multicomponent multidisciplinary bundle of interventions on sleep and delirium in medical and surgical intensive care patients. Anaesthesia. 2014 Jun;69(6):540-9. doi: 10.1111/anae.12638. PMID 24813132
- [Background] Pulak LM, Jensen L. Sleep in the Intensive Care Unit: A Review. J Intensive Care Med. 2016 Jan;31(1):14-23. doi: 10.1177/0885066614538749. Epub 2014 Jun 10. PMID 24916753
- [Background] Ritmala-Castren M, Virtanen I, Leivo S, Kaukonen KM, Leino-Kilpi H. Sleep and nursing care activities in an intensive care unit. Nurs Health Sci. 2015 Sep;17(3):354-61. doi: 10.1111/nhs.12195. Epub 2015 Mar 18. PMID 25786544
- [Background] Weinhouse GL, Schwab RJ. Sleep in the critically ill patient. Sleep. 2006 May;29(5):707-16. doi: 10.1093/sleep/29.5.707. PMID 16774162
- [Background] White BL, Zomorodi M. Perceived and actual noise levels in critical care units. Intensive Crit Care Nurs. 2017 Feb;38:18-23. doi: 10.1016/j.iccn.2016.06.004. Epub 2016 Aug 25. PMID 27567305
- [Derived] Tonna JE, Dalton A, Presson AP, Zhang C, Colantuoni E, Lander K, Howard S, Beynon J, Kamdar BB. The Effect of a Quality Improvement Intervention on Sleep and Delirium in Critically Ill Patients in a Surgical ICU. Chest. 2021 Sep;160(3):899-908. doi: 10.1016/j.chest.2021.03.030. Epub 2021 Mar 24. PMID 33773988